CLINICAL TRIAL: NCT03904316
Title: Use of Biodesign® Otologic Graft in Tympanoplasty: A Prospective, Randomized Trial
Brief Title: Use of Biodesign® Otologic Graft in Tympanoplasty
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: The trial was stopped as the benefit was challenging to determine in preliminary usage.
Sponsor: Henry Ford Health System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1322227
Record Dates: First submitted 2019-03-18; First posted 2019-04-05 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2022-08

CONDITIONS: Tympanic Membrane Perforation
MeSH Terms: conditions — Tympanic Membrane Perforation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Biodesign graft tympanic membrane repair (Experimental): Patient's perforated tympanic membrane will be repaired with an acellular matrix derived from porcine small intestine submucosa, Biodesign Otologic graft
  Interventions: Biological: Biodesign Otologic graft
- Autograft tympanic membrane repair (Active Comparator): Patient's perforated tympanic membrane will be repaired with autologous temporalis fascia.
  Interventions: Other: Autologous temporalis fascia

INTERVENTIONS:
Biological: Biodesign Otologic graft — Acellular matrix derived from porcine small intestine submucosa
  Arms: Biodesign graft tympanic membrane repair
Other: Autologous temporalis fascia — An autologous graft for tympanic membrane repair
  Arms: Autograft tympanic membrane repair

SUMMARY:
This is a prospective, randomized trial to evaluate tympanoplasty outcomes using Biodesign SIS graft compared to autologous temporalis fascia, the most commonly used graft for repair of tympanic membrane.

DETAILED DESCRIPTION:
Patients 18 years or older will undergo primary tympanoplasty without mastoidectomy. The patients will be randomized into groups receiving Biodesign versus autograft temporalis fascia for repair.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing primary tympanoplasty without mastoidectomy.

Exclusion Criteria:

* Patients with a known biologic sensitivity or a cultural objection to use of porcine materials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-10-03 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Assessment of graft take after tympanoplasty | 1 month postoperatively by the surgeon
  Microscopically evaluate tympanic membrane for perforation closure
Assessment of graft take after tympanoplasty | 2 months postoperatively by the surgeon
  Microscopically evaluate tympanic membrane for perforation closure
Assessment of graft take after tympanoplasty | 3 months postoperatively by the surgeon
  Microscopically evaluate tympanic membrane for perforation closure
Assessment of graft take after tympanoplasty | 6 months postoperatively by the surgeon
  Microscopically evaluate tympanic membrane for perforation closure

SECONDARY OUTCOMES:
Measurement of Hearing Parameters | Measure hearing parameters preoperatively
  Test the pure tone conduction (average of 500, 1000 and 2000 Hz).
Measurement of Hearing Parameters | Measure hearing parameters preoperatively.
  Test the Air Bone Gap starting at 1000 Hz then 2000, 4000, 8000, 250 and 500 for air-conduction thresholds. Then test non-masked bone-conduction thresholds at the same frequencies.
Measurement of Hearing Parameters | Measure hearing parameters preoperatively
  Test Word Recognition for 50-2 syllables words
Measurement of Hearing Parameters | Measure hearing parameters 3 months postoperatively
  Test the pure tone conduction (average of 500, 1000 and 2000 Hz).
Measurement of Hearing Parameters | Measure hearing parameters 3 months postoperatively
  Determine the air bond gap by measuring the difference between the air conduction and gone conduction testing. The air bone gap is the difference between the 2 readings and must be present at 3 consecutive frequencies.
Measurement of Hearing Parameters | Measure hearing parameters 3 months postoperatively
  The word recognition testing evaluates the patient's ability to repeat phonetically balanced words appropriate for his/her hearing level.
Measurement of Hearing Parameters | Measure hearing parameters 6 months postoperatively
  Test the pure tone conduction (average of 500, 1000 and 2000 Hz).
Measurement of Hearing Parameters | Measure hearing parameters 6 months postoperatively
  Determine the air bond gap by measuring the difference between the air conduction and gone conduction testing. The air bone gap is the difference between the 2 readings and must be present at 3 consecutive frequencies.
Measurement of Hearing Parameters | Measure hearing parameters 6 months postoperatively
  The word recognition testing evaluates the patient's ability to repeat phonetically balanced words appropriate for his/her hearing level.

CONTACTS AND LOCATIONS:
Overall Officials: Seilesh Babu, MD, Principal Investigator — Michigan Ear Institute
Locations (1):
- Ascension Providence Hospital, Novi Campus, Novi, Michigan, United States

REFERENCES:
- [Background] Ambro BT, Zimmerman J, Rosenthal M, Pribitkin EA. Nasal septal perforation repair with porcine small intestinal submucosa. Arch Facial Plast Surg. 2003 Nov-Dec;5(6):528-9. doi: 10.1001/archfaci.5.6.528. PMID 14623693
- [Background] Ansaloni L, Cambrini P, Catena F, Di Saverio S, Gagliardi S, Gazzotti F, Hodde JP, Metzger DW, D'Alessandro L, Pinna AD. Immune response to small intestinal submucosa (surgisis) implant in humans: preliminary observations. J Invest Surg. 2007 Jul-Aug;20(4):237-41. doi: 10.1080/08941930701481296. PMID 17710604
- [Background] Bejjani GK, Zabramski J; Durasis Study Group. Safety and efficacy of the porcine small intestinal submucosa dural substitute: results of a prospective multicenter study and literature review. J Neurosurg. 2007 Jun;106(6):1028-33. doi: 10.3171/jns.2007.106.6.1028. PMID 17564175
- [Background] Illing E, Chaaban MR, Riley KO, Woodworth BA. Porcine small intestine submucosal graft for endoscopic skull base reconstruction. Int Forum Allergy Rhinol. 2013 Nov;3(11):928-32. doi: 10.1002/alr.21206. Epub 2013 Aug 16. PMID 23956139
- [Background] JANSEN C. CARTILAGE--TYMPANOPLASTY. Laryngoscope. 1963 Oct;73:1288-301. doi: 10.1288/00005537-196310000-00006. No abstract available. PMID 14073760
- [Background] Knoll LD. Use of porcine small intestinal submucosal graft in the surgical management of Peyronie's disease. Urology. 2001 Apr;57(4):753-7. doi: 10.1016/s0090-4295(00)01079-7. PMID 11306396
- [Background] Lin HK, Godiwalla SY, Palmer B, Frimberger D, Yang Q, Madihally SV, Fung KM, Kropp BP. Understanding roles of porcine small intestinal submucosa in urinary bladder regeneration: identification of variable regenerative characteristics of small intestinal submucosa. Tissue Eng Part B Rev. 2014 Feb;20(1):73-83. doi: 10.1089/ten.TEB.2013.0126. Epub 2013 Jul 25. PMID 23777420
- [Background] Min J, Kim SH. Comparison of transcanal endoscopic tympanoplasty with sterile acellular dermal allograft to conventional endaural microscopic tympanoplasty with tragal perichondrium. Am J Otolaryngol. 2018 Mar-Apr;39(2):167-170. doi: 10.1016/j.amjoto.2017.11.014. Epub 2017 Dec 7. PMID 29290312
- [Background] Murphy F, Corbally MT. The novel use of small intestinal submucosal matrix for chest wall reconstruction following Ewing's tumour resection. Pediatr Surg Int. 2007 Apr;23(4):353-6. doi: 10.1007/s00383-007-1882-1. Epub 2007 Feb 8. PMID 17287942
- [Background] Ort SA, Ehrlich HP, Isaacson JE. Acellular porcine intestinal submucosa as fascial graft in an animal model: applications for revision tympanoplasty. Otolaryngol Head Neck Surg. 2010 Sep;143(3):435-40. doi: 10.1016/j.otohns.2010.04.268. PMID 20723784
- [Background] ORTEGREN U. MYRINGOPLASTY. A 4-YEAR SERIES REVIEWED 2 YEARS AFTER OPERATION. Acta Otolaryngol Suppl. 1964;188:SUPPL 188:234+. No abstract available. PMID 14146678
- [Background] Phillips J, Riley KO, Woodworth BA. Porcine small intestine submucosal grafts for post-tumor resection orbital reconstruction. Laryngoscope. 2014 Jun;124(6):E219-23. doi: 10.1002/lary.24515. Epub 2013 Dec 18. PMID 24214917
- [Background] Van Rompaey V, Farr MR, Hamans E, Mudry A, Van de Heyning PH. Allograft tympanoplasty: a historical perspective. Otol Neurotol. 2013 Jan;34(1):180-8. doi: 10.1097/MAO.0b013e31826bf16d. PMID 23032665
- [Background] Rutner AB, Levine SR, Schmaelzle JF. Processed porcine small intestine submucosa as a graft material for pubovaginal slings: durability and results. Urology. 2003 Nov;62(5):805-9. doi: 10.1016/s0090-4295(03)00664-2. PMID 14624898
- [Background] Seymour PE, Leventhal DD, Pribitkin EA. Lip augmentation with porcine small intestinal submucosa. Arch Facial Plast Surg. 2008 Jan-Feb;10(1):30-3. doi: 10.1001/archfacial.2007.17. PMID 18209120
- [Background] SHEA JJ Jr. Vein graft closure of eardrum perforations. J Laryngol Otol. 1960 Jun;74:358-62. doi: 10.1017/s002221510005670x. No abstract available. PMID 13854782
- [Background] Spiegel JH, Kessler JL. Tympanic membrane perforation repair with acellular porcine submucosa. Otol Neurotol. 2005 Jul;26(4):563-6. doi: 10.1097/01.mao.0000169636.63440.4e. PMID 16015147
- [Background] Storrs L. Myringoplasty. Laryngoscope. 1966 Feb;76(2):185-95. doi: 10.1288/00005537-196602000-00001. No abstract available. PMID 5324120
- [Background] Tan HE, Santa Maria PL, Eikelboom RH, Anandacoomaraswamy KS, Atlas MD. Type I Tympanoplasty Meta-Analysis: A Single Variable Analysis. Otol Neurotol. 2016 Aug;37(7):838-46. doi: 10.1097/MAO.0000000000001099. PMID 27273405